CLINICAL TRIAL: NCT02873741
Title: New Strategies to Assess Anal Cancer Risk In Women
Acronym: ANCAR-WIHS
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Lisa Flowers, Professor, Emory University
Other Study IDs: IRB00083800; U01AI103408-03 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-19 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Human Immunodeficiency Virus (HIV); Human Papillomavirus (HPV)
Keywords: Sexually Transmitted Diseases (STDs); Cancer; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validation Study: Participants will undergo a perianal and digital anorectal exam, a high resolution anoscopy, and cervical and anal swabs to determine the best method to identify women at high risk for anal cancer.
  Interventions: Procedure: Perianal and Digital Anorectal Exam; Procedure: Cervical Swabs; Procedure: Anal Swabs; Procedure: High Resolution Anoscopy (HRA)

INTERVENTIONS:
Procedure: Perianal and Digital Anorectal Exam — The physician will inspect the outside of the anus and use a gloved finger to feel the anus for any masses.
Procedure: Cervical Swabs — A speculum will be inserted into the vagina to visualize the cervix. The sample for research tests will be collected with one ThinPrep cytobroom inserted into the cervix. Collection will be same for the sample to be paced in the RNA storage solution for future biomarker studies.
Procedure: Anal Swabs — The anal cytology specimen will be collected by inserting a saline moistened cotton-tipped swab into the anus, rotating it clock-wise for 20 seconds, and placed in SurePath. The first twenty participants will have anal cells collected in two different ways for validation/optimization: 1) saline moistened Dacron swab placed directly in ThinPrep medium and 2) Medscand Cytobrush Plus, a special brush, placed directly into ThinPrep medium. After validation/optimization is complete for up to 20 participants, the best collection method will be selected and will be used for all future enrolled participants.
Procedure: High Resolution Anoscopy (HRA) — High Resolution Anoscopy is a procedure that allows for examination and evaluation of the anal canal. Using a small thin round tube called an anoscope, the anal canal is examined with a high resolution magnifying instrument called a colposcope. Application of a mild acidic liquid (acetic acid or diluted vinegar) or a brown iodine-based solution (Lugol's) onto the anal canal facilitates evaluation of abnormal tissue such as anal dysplasia. If abnormal staining is seen using acetic acid (dense white lesion) or Lugol's solution (bright yellow lesion) a biopsy of that area will be obtained.

SUMMARY:
The purpose of this research is to study different strategies to identify women at highest risk for anal cancer. Primarily, investigators want to study a risk assessment called the Anal Cancer Risk Index; it gives women an overall number score based on risk factors that they may have for anal cancer, such as age, number of sexual partners, or smoking. Investigators seek to understand whether women with higher Anal Cancer Risk Index scores are more likely to have abnormal results on anal pap smears, HPV tests, or anal biopsies. The study team will collect swabs of the cervix and the anus to study different laboratory tests that could identify women at highest risk of cervical and anal cancer. These laboratory tests include an anal pap smear, tests for markers of disease and tests that detect the HPV types most likely to cause cancer. The study team would like to see which of these laboratory tests do the best job at predicting precancerous lesions in the anus and are better indicators of risk for cancer. After collecting these swabs, women will have a procedure called high resolution anoscopy where investigators look closely at the anus and biopsy any suspicious areas. Finally, the study team will look for HPV proteins and changes that HPV can make in cells to see if these tests predict anal lesions.

DETAILED DESCRIPTION:
Investigators seek to study different strategies to identify women at highest risk for anal cancer. Primarily, investigators want to study a risk assessment called the Anal Cancer Risk Index; it gives women an overall number score based on risk factors that they may have for anal cancer, such as age, number of sexual partners, or smoking. The study team would like to determine whether women with higher Anal Cancer Risk Index scores are more likely to have abnormal results on anal pap smears, HPV tests, or anal biopsies. Next, the team will collect a swab of the cervix and swabs of the anus to study different laboratory tests that could identify women at highest risk of anal cancer: these tests include an anal pap smear and tests that detect HPV types most likely to cause cancer. Investigators would like to see which of these laboratory tests do the best job at predicting precancerous lesions in the anus. After collecting these swabs, women will have a procedure called high resolution anoscopy where investigators will look closely at the anus and biopsy any suspicious areas. Finally, the study team will look for HPV proteins and changes that HPV can make in cells to see if these tests predict anal lesions. The HPV protein is called E6 and E7 and the cell change test is called CADM1/MAL/miR-124-2. Investigators will measure E6/E7 and CADM1/MAL/miR-124-2 in cervical and anal samples to see if women positive for this marker are more likely to have abnormal results on anal pap smears or anal biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in the Women's HIV Interagency Study (WIHS) study
* Able and willing to undergo anal cytology, anal molecular testing, and high resolution anoscopy with targeted anal biopsies

Exclusion Criteria:

* History of high grade anal intraepithelial neoplasia (AIN 2 or 3)
* History of active anal disease requiring surgery
* History of anal or cervical cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women enrolled in the Atlanta WIHS without history of high grade AIN or anal cancer will be eligible to enroll in this study and will be contacted by a research coordinator.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2016-07; Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Anal Cancer Risk Index Score | Day 1
  Assessment of anal cancer screening, risk factors for anal cancer, and its association with HPV using AIDS Risk Reduction Model Framework, that is a three stage model, including knowledge as a prerequisite to recognize risk and to take action to change or reduce the risk. Knowledge was measured with the Knowledge of Anal cancer and HPV, that is a 44-item knowledge multiple choice survey adapted from the Hild-Mosely, et al study, substituting "cervical" with "anal". A percentage score of correct responses was calculated and range from o to 100, being 100 the maximum correct result.
Presence of Anal hr-HPV | Day 1
  Assessment of high risk human papilloma virus in the anal cytology.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Flowers, MD, Principal Investigator — Emory University
Locations (1):
- The Ponce Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wells JS, Flowers L, Paul S, Nguyen ML, Sharma A, Holstad M. Knowledge of Anal Cancer, Anal Cancer Screening, and HPV in HIV-Positive and High-Risk HIV-Negative Women. J Cancer Educ. 2020 Jun;35(3):606-615. doi: 10.1007/s13187-019-01503-8. PMID 30850945
- [Background] Lahiri CD, Nguyen ML, Mehta CC, Mosunjac M, Tadros T, Unger ER, Rajeevan MS, Richards J, Ofotokun I, Flowers L. Pilot Study of Markers for High-grade Anal Dysplasia in a Southern Cohort From the Women's Interagency Human Immunodeficiency Virus Study. Clin Infect Dis. 2020 Mar 3;70(6):1121-1128. doi: 10.1093/cid/ciz336. PMID 31058984